CLINICAL TRIAL: NCT06497465
Title: Dolutegravir Plus Lamivudine (DTG/3TC) Dual Therapy Versus Dolutegravir With TDF-lamivudine (DTG + TDF/3TC) Among Antiretroviral naïve People With HIV and TB Receiving Rifampin-based TB Treatment
Brief Title: Dolutegravir/Lamivudine Dual Therapy for ART-naïve People With HIV and TB Receiving Rifampin-based TB Treatment
Acronym: DOVETAIL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00441778
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis; HIV
MeSH Terms: conditions — Tuberculosis | interventions — dolutegravir; Lamivudine; Tenofovir

STUDY DESIGN:
Intervention Model Description: Arm 1(n=50): DTG 50mg/3TC 300 mg FDC tablet (Dovato®) twice daily during TB therapy and for 2 weeks after, then Dolutegravir (DTG) 50mg / lamivudine (3TC) 300 mg fixed dose combination (FDC) tablet (Dovato®) once daily to week 52
  Arm 2(n=50): DTG 50mg/300mg FDC tablet plus DTG 50mg at night during TB treatment and for 2 weeks after, then DTG 50 mg/ 3TC 300 mg FDC tablet (Dovato®) once daily to week 52
  Arm 3(n=50): Local Standard of Care 3-drug ART (DTG 50mg + TDF/3TC) plus DTG 50 mg at night during TB treatment and for 2 weeks after, then Dolutegravir (DTG) 50 mg + Tenofovir disoproxil fumarate (TDF)/ lamivudine (3TC) FDC tablet once daily to week 52
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: DTG 50 mg/ 3TC 300mg (Dovato®) twice daily (BID) (Experimental): Arm 1: DTG 50mg/3TC 300 mg fixed-dose-combination (FDC) tablet (Dovato®) twice daily during TB therapy and for 2 weeks after, then DTG 50mg/3TC 300 mg FDC tablet (Dovato®) once daily to week 52
  Interventions: Drug: Dolutegravir/Lamivudine 50 MG-300mg Oral Tablet [DOVATO]
- Arm 2: DTG 50 mg/ 3TC 300mg (Dovato®) once daily (QD) in the morning with DTG 50 mg in the evening (Experimental): Arm 2: DTG 50mg/300mg FDC tablet plus DTG 50mg at night during TB treatment and for 2 weeks after, then DTG 50 mg/ 3TC 300 mg FDC tablet (Dovato®) once daily to week 52
  Interventions: Drug: Dolutegravir 50mg Tab; Drug: Dolutegravir/Lamivudine 50 MG-300mg Oral Tablet [DOVATO]
- Arm 3: Standard of Care 3-drug ART (DTG+ TDF/3TC) plus DTG 50mg in the evening. (Active Comparator): Arm 3: Local Standard of Care 3-drug ART (DTG 50mg + TDF/3TC) plus DTG 50 mg at night during TB treatment and for 2 weeks after, then DTG 50 mg + TDF/3TC FDC tablet once daily to week 52
  Interventions: Drug: Dolutegravir plus Tenofovir disoproxil fumarate (TDF)/ lamivudine (3TC)

INTERVENTIONS:
Drug: Dolutegravir 50mg Tab — Participants will receive Dolutegravir 50mg
  Other Names: TIVICAY 50 mg; TIVICAY PD
  Arms: Arm 2: DTG 50 mg/ 3TC 300mg (Dovato®) once daily (QD) in the morning with DTG 50 mg in the evening
Drug: Dolutegravir/Lamivudine 50 MG-300mg Oral Tablet [DOVATO] — Participants will receive Dolutegravir/Lamivudine 50 MG-300 MG Oral Tablet [DOVATO]
  Arms: Arm 1: DTG 50 mg/ 3TC 300mg (Dovato®) twice daily (BID); Arm 2: DTG 50 mg/ 3TC 300mg (Dovato®) once daily (QD) in the morning with DTG 50 mg in the evening
Drug: Dolutegravir plus Tenofovir disoproxil fumarate (TDF)/ lamivudine (3TC) — Participants will receive Dolutegravir plus Tenofovir disoproxil fumarate (TDF)/ lamivudine (3TC)
  Arms: Arm 3: Standard of Care 3-drug ART (DTG+ TDF/3TC) plus DTG 50mg in the evening.

SUMMARY:
This will be a Phase IIIb Clinical Trial, an international multicenter, randomized, three-arm, non-comparative trial of efficacy, safety, and tolerability of the dual therapy regimen dolutegravir plus lamivudine either twice daily or DTG/3TC ( Dovato) in the morning +dolutegravir (DTG) in the evening, versus standard of care (SOC) twice-daily dolutegravir plus 2 once-daily Nucleoside reverse-transcriptase inhibitors (NRTIs) tenofovir disoproxil fumarate /lamivudine (TDF/3TC), among antiretroviral therapy (ART)-nave individuals with HIV-1 receiving rifampin-based TB therapy

DETAILED DESCRIPTION:
Tuberculosis (TB) is the most common cause of death in people with HIV worldwide. Among patients with HIV, the incidence of TB per year is about 5-10%. The two diseases are now always treated concurrently in co-infected individuals, as there is a survival benefit for starting antiretroviral therapy (ART) soon after TB treatment initiation. Current Brazilian guidelines suggest that for patients with a cluster of differentiation 4 (CD4) < 50, ART should be started within 2 weeks of starting TB treatment; for patients with a CD4>50, ART should be started within 2 months of starting TB treatment. World Health Organization guidelines suggest ART initiation within 2 weeks of TB diagnosis regardless of CD4 count (provided there are no signs of TB meningitis), but most programs defer ART until 6-8 weeks in patients with CD4 >50 to reduce the risk of immune reconstitution inflammatory syndrome (IRIS).

The option of dual therapy for HIV (i.e., complete regimens to treat HIV composed of only 2 drugs) is of increasing interest and can lower costs for patients, payors, and programs while lowering cumulative lifetime exposure to ART (with potential resultant lessened burden of cumulative toxicities) and maintaining high antiviral efficacy. Based on the GEMINI, TANGO, and SALSA clinical trials, a regimen of 50 milligram (mg) DTG combined with 300mg lamivudine (3TC) has been shown to be a highly effective stand-alone option for the treatment of HIV-1 in ART treatment-naïve or virologically suppressed individuals through 48 weeks (SALSA) and 144 weeks (GEMINI and TANGO).

ELIGIBILITY:
Inclusion Criteria:

* Documentation of HIV-1 status: HIV-1 infection, documented by any licensed rapid HIV test or HIV-1 enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, or plasma HIV 1 RNA viral load. Two or more HIV-1 RNA viral loads of >1,000 copies/mL are also acceptable as documentation of HIV-1 infection.
* CD4+ cell count ≥50 cells/mm3 obtained within 30 days prior to study entry
* HIV-1 viral load ≥1000 copies/mL
* ART-naïve.
* Documentation of pulmonary TB

Exclusion Criteria:

* Pregnant, or plans to become pregnant.

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Among treatment-naïve participants with HIV-1 who are taking rifampin-based regimens for TB, determine the proportion with HIV-1 virologic suppression (via FDA snapshot algorithm) at 28 weeks of HIV treatment, by arm | 28 weeks
  To Compare the proportion of participants with HIV-1 virologic suppression at 28 weeks of HIV treatment by arm.

SECONDARY OUTCOMES:
1.3.1 Number of patients with HIV-1 virologic suppression (via FDA snapshot algorithm) at 48 weeks, in each arm | 48 weeks
  To compare the proportion in each arm above DTG protein adjusted 90% inhibitory concentration (IC90) (64 ng/mL) at each PK sampling.
1.3.2 Number of patients with HIV-1 virologic suppression at 48 weeks, in the combined DTG/3TC arms (Arm 1 + Arm 2) | 48 weeks
  To compare the proportion of patients with HIV-1 virologic suppression at 48 weeks, in the combined DTG/3TC arms (Arm 1 + Arm 2)
1.3.3 Change from baseline in CD4 over 28 weeks and 48 weeks of HIV treatment, by arm | 28 weeks, 48 weeks
  To compare the changes from baseline over 28 weeks and 48 weeks of HIV treatment by the arm.
1.3.4 Proportion of participants with DTG Cmin above target DTG trough of 158 ng/mL | 2years
  1-To estimate the pharmacokinetics (PK) of DTG when given twice daily as a 50 mg/ 300 mg DTG/3TC FDC with rifampicin (RIF)-containing TB treatment, X DTG 50 mg/ 3TC 300 mg FDC given once daily without RIF among the same participants after completing TB treatment.
1.3.4 Concentration of the PK of DTG | 2years
  Concentration of DTG when given twice daily as a 50 mg/ 300 mg DTG/3TC FDC with RIF-containing TB treatment, X DTG 50 mg/ 3TC 300 mg FDC given once daily without RIF among the same participants after completing TB treatment.
1.3.5 Compare Grade 3 or 4 adverse events, by arm | 2 years
  To compare the Grade 3 & 4 adverse events by arm

CONTACTS AND LOCATIONS:
Overall Officials: Ethel M Weld, MD, Principal Investigator — Johns Hopkins University
Locations (6):
- Brazil (6):
  - Instituto Tropical de Doenças Infecciosas Manaus, Manaus, Amazonas
  - Universidade Federal da Bahia, Salvador, Estado de Bahia
  - FIOCruz, Rio de Janeiro, Rio de Janeiro
  - Hospital Geral de Nova Iguaçu, Rio de Janeiro, Rio de Janeiro
  - CePClin - Center for Studies and Research in Infectious Diseases Ltda, Natal, Rio Grande do Norte
  - RDSS- Ricardo Diaz Solucoes Cientificas, São Paulo, São Paulo